CLINICAL TRIAL: NCT04449679
Title: Real-Time Monitoring of Chemotherapy Side Effects in Patients With Gastro-Intestinal Malignancies
Brief Title: Real-Time Monitoring of Chemotherapy Side-Effects in Patients With Gastrointestinal Cancers, RT-CAMSS Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20G.090; JT 15039 (Other: JeffTrial Number)
Record Dates: First submitted 2020-05-13; First posted 2020-06-29 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Clinical Stage 0 Esophageal Adenocarcinoma AJCC v8; Clinical Stage 0 Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage 0 Gastric Cancer AJCC v8; Clinical Stage I Esophageal Adenocarcinoma AJCC v8; Clinical Stage I Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage I Gastric Cancer AJCC v8; Clinical Stage II Esophageal Adenocarcinoma AJCC v8; Clinical Stage II Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage II Gastric Cancer AJCC v8; Clinical Stage IIA Esophageal Adenocarcinoma AJCC v8; Clinical Stage IIA Gastric Cancer AJCC v8; Clinical Stage IIB Gastric Cancer AJCC v8; Clinical Stage III Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage III Gastric Cancer AJCC v8; Clinical Stage IV Esophageal Adenocarcinoma AJCC v8; Clinical Stage IV Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IV Gastric Cancer AJCC v8; Clinical Stage IVA Esophageal Adenocarcinoma AJCC v8; Clinical Stage IVA Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IVA Gastric Cancer AJCC v8; Clinical Stage IVB Esophageal Adenocarcinoma AJCC v8; Clinical Stage IVB Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IVB Gastric Cancer AJCC v8; Pathologic Stage 0 Esophageal Adenocarcinoma AJCC v8; Pathologic Stage 0 Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage 0 Gastric Cancer AJCC v8; Pathologic Stage I Esophageal Adenocarcinoma AJCC v8; Pathologic Stage I Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage I Gastric Cancer AJCC v8; Pathologic Stage IA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IA Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IA Gastric Cancer AJCC v8; Pathologic Stage IB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IB Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IB Gastric Cancer AJCC v8; Pathologic Stage IC Esophageal Adenocarcinoma AJCC v8; Pathologic Stage II Esophageal Adenocarcinoma AJCC v8; Pathologic Stage II Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage II Gastric Cancer AJCC v8; Pathologic Stage IIA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIA Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IIA Gastric Cancer AJCC v8; Pathologic Stage IIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIB Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IIB Gastric Cancer AJCC v8; Pathologic Stage III Esophageal Adenocarcinoma AJCC v8; Pathologic Stage III Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage III Gastric Cancer AJCC v8; Pathologic Stage IIIA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIA Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IIIA Gastric Cancer AJCC v8; Pathologic Stage IIIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIB Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IIIB Gastric Cancer AJCC v8; Pathologic Stage IIIC Gastric Cancer AJCC v8; Pathologic Stage IV Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IV Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IV Gastric Cancer AJCC v8; Pathologic Stage IVA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IVA Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IVB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IVB Esophageal Squamous Cell Carcinoma AJCC v8; Stage 0 Colorectal Cancer AJCC v8; Stage 0 Pancreatic Cancer AJCC v8; Stage I Colorectal Cancer AJCC v8; Stage I Pancreatic Cancer AJCC v8; Stage IA Pancreatic Cancer AJCC v8; Stage IB Pancreatic Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage II Pancreatic Cancer AJCC v8; Stage IIA Colorectal Cancer AJCC v8; Stage IIA Pancreatic Cancer AJCC v8; Stage IIB Colorectal Cancer AJCC v8; Stage IIB Pancreatic Cancer AJCC v8; Stage IIC Colorectal Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms | interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: PHASE I: Patients participate in an audio-recorded focus group or one-on-one interview over 40 minutes either in-person, over the phone, or electronically. Patients receive sample text messages and questionnaires generated from the RT-CAMSS to generate reaction, discussion, and scenarios.
  PHASE II: Patients receive RT-CAMSS over 2 months or until chemotherapy is discontinued, whichever is earlier. RT-CAMSS consists of text messages addressing knowledge about specific cancer type and chemotherapy, side-effect prevention, suggestions of lifestyle behavioral changes and emotional support, and preparation for surgery. Patients then record their symptoms through answering a series of questionnaires and receive tailored feedback according to their answers, including a consultation with a nurse.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Services Research (RT-CAMSS) (Experimental): Patients receive RT-CAMSS over 2 months or until chemotherapy is discontinued, whichever is earlier. RT-CAMSS consists of text messages addressing knowledge about specific cancer type and chemotherapy, side-effect prevention, suggestions of lifestyle behavioral changes and emotional support, and preparation for surgery. Patients then record their symptoms through answering a series of questionnaires and receive tailored feedback according to their answers, including a consultation with a nurse.
  Interventions: Other: Patient Monitoring System; Other: Questionnaire Administration; Other: Consultation

INTERVENTIONS:
Other: Patient Monitoring System — Receive RT-CAMSS
Other: Questionnaire Administration — Complete questionnaires
Other: Consultation — Receive tailored feedback, including consultation with nurse
  Other Names: Consult

SUMMARY:
This trial tests new methods and materials for the real-time chemotherapy-associated side effects monitoring support system (RT-CAMSS) in patients with gastrointestinal cancers undergoing chemotherapy. RT-CAMSS is a monitoring support system that provides patients with evidence-based information and side-effect management and coping skills, emotional support and validation, and proactive care via text messages and questionnaires as they undergo chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop and refine a real-time chemo-associated side effects monitoring support system (RT-CAMSS) using interactive text messaging (TXT) for patients with gastric, esophageal, pancreatic and colorectal cancer during chemotherapy.

II. Assess the feasibility and engagement of the RT-CAMSS in a 2-month pilot study.

III. To gather preliminary data on the impact of RT-CAMSS on patient's quality of life and symptom distress.

OUTLINE:

PHASE I: Patients participate in an audio-recorded focus group or one-on-one interview over 40 minutes either in-person, over the phone, or electronically. Patients receive sample text messages and questionnaires generated from the RT-CAMSS to generate reaction, discussion, and scenarios.

PHASE II: Patients receive RT-CAMSS over 2 months or until chemotherapy is discontinued, whichever is earlier. RT-CAMSS consists of text messages addressing knowledge about specific cancer type and chemotherapy, side-effect prevention, suggestions of lifestyle behavioral changes and emotional support, and preparation for surgery. Patients then record their symptoms through answering a series of questionnaires and receive tailored feedback according to their answers, including a consultation with a nurse.

After completion of study, patients are followed up at 1 and 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with gastric, esophageal, pancreatic or colorectal cancer
* Scheduled to start intravenous (IV) chemotherapy or has started IV chemotherapy
* Able to read and understand English
* Able to provide signed and dated informed consent form
* Have a mobile device with text message capability
* Know or willing to learn how to use text messaging

Exclusion Criteria:

* < 18 years of age
* Cognitive impairment documented in the electronic medical record (EMR), biological variables (sex)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Feasibility and Engagement | Up to 2 months or until chemotherapy is discontinued, whichever is earlier
  Will be measured through study accrual, attrition, and system usage frequencies. We aim for accrual at a rate of 50% to match our prior study but a rate over 30% will be feasible. The intervention will be considered feasible if attrition does not exceed 30%. 90% of participants reporting their symptoms at least once will be considered adequate.
Acceptability | Up to 2 months or until chemotherapy is discontinued, whichever is earlier
  Will be measured through a satisfaction measure and patient interview data. Acceptability will be established by a group median score >= 3 on the 1-4 satisfaction scale.
Symptom distress | Up to 2 months or until chemotherapy is discontinued, whichever is earlier
  The Memorial Symptom Assessment Scale (MSAS), a well-validated instrument that will be used to assess common physical symptoms concerning chemotherapy in patients. The MSAS measures the prevalence, frequency, severity, and distress of 25 physical symptoms and seven psychological symptoms.
Self-efficacy | Up to 2 months or until chemotherapy is discontinued, whichever is earlier
  Will be measured using the Patient Activation Measure (PAM) for assessing skills, knowledge and self-confidence for self-management. The scale asks participants concerning their certainty of controlling symptoms caused by chemotherapy to perform daily activities.
Information and support needs | Prior to start of chemotherapy treatment
  Will be measured using the Cancer Treatment Scale (CaTS). The CaTS assesses patient's preparation prior to the start of their chemotherapy treatment.
Medical information | Baseline
  Will be extracted from the electronic medical record (EMR) chart including cancer diagnosis information, treatment schedule and discontinuation.
Functional Assessment of Cancer Treatment - General scale | Up to 2 months or until chemotherapy is discontinued, whichever is earlier
  Questionnaire will be used to assess patient quality of life. The 27-item FACT-G assesses four specific domains including physical, social, emotional and functional well-being.
Social support | Up to 2 months or until chemotherapy is discontinued, whichever is earlier
  The Multidemensional Scale of Perceived Social Support (MSPSS), a well-validated 12-item instrument used to assess patient perceived social support.
Post-intervention evaluation | Through study completion, an average of 2 months
  Patient interviews will explore key domains including perceived usefulness, how well the enhanced usual care and the RT-CAMSS address their concerns, whether there are additional issues they would like to see included and the characteristics of the text message.

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-Yi Wen, MD, Principal Investigator — Thomas Jefferson University Hospital, Philadelphia, PA 19107 USA
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States